CLINICAL TRIAL: NCT01755091
Title: Cannabimimetic Treatment of Obstructive Sleep Apnea: A Proof of Concept Trial
Brief Title: Safety and Efficacy Study of Dronabinol to Treat Obstructive Sleep Apnea
Acronym: PACE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Northwestern University (Other); University of Chicago (Other); Hektoen Institute for Medical Research (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, David W. Carley, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012-0095; UM1HL112856 (NIH)
Record Dates: First submitted 2012-12-18; First posted 2012-12-21 (Estimated); Results first posted 2017-12-22 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sugar Pill (Placebo Comparator): Placebo, once per day (QD) by mouth, 60 minutes before bedtime for 6 weeks after 1-week run-in
  Interventions: Drug: Placebo (for Dronabinol)
- 2.5 mg/day (Experimental): Dronabinol, 2.5 mg QD by mouth, 60 minutes before bedtime for 6 weeks after 1-week placebo run-in
  Interventions: Drug: Dronabinol
- 10 mg/day (Experimental): Dronabinol, 10 mg QD by mouth, 60 minutes before bedtime for 4 weeks after 1-week placebo run-in and 2-week dose escalation
  Interventions: Drug: Dronabinol

INTERVENTIONS:
Drug: Dronabinol
  Arms: 10 mg/day; 2.5 mg/day
Drug: Placebo (for Dronabinol)
  Arms: Sugar Pill

SUMMARY:
This is a proof of concept study to determine the safety and efficacy of dronabinol for the treatment of obstructive sleep apnea syndrome (OSA).

ELIGIBILITY:
Inclusion Criteria:

* Adult 21 to 64 years of age;
* 15≤AHI ≤ 50 on screening polysomnogram (PSG)
* ESS score ≥ 7
* Able to understand and complete informed consent and all study assessments and forms, presented in an English-speaking format;
* Women of child-bearing potential (WCBP) must have a negative urine pregnancy test. In addition sexually active WCBP must agree to use adequate contraceptive methods (oral, injectable or implantable hormonal contraceptive; tubal ligation; intra-uterine devices; barrier contraceptive with spermicide; or vasectomized partner).

Exclusion Criteria:

* Arterial oxygen saturation < 75% for > 5% of sleep period time on screening PSG;
* Occupation or life situation that may impart risk by study participation (e.g. commercial driver, pilot, police officer, fireman);
* Motor vehicle accident or "near-miss" related to sleepiness (self-report) within 2 years of the first dose of study drug (Day 8);
* Body mass index > 45 kg/m2
* Severe obstructive sleep apnea syndrome (OSAS) that, based on the clinical judgment of the Investigator, precludes delaying positive airway pressure treatment;
* History of shift work or rotating shifts within the month prior to the first dose of study drug (Day 8);
* Prior upper airway surgery for snoring or OSAS as an adult (≥ 18 years of age);
* Prior non-invasive treatment for OSAS within 6 months prior to the first dose of study drug (Day 8);
* Major surgery within 6 months prior to the first dose of study drug (Day 8);
* Bariatric surgery within 2 years prior to the first dose of study drug (Day 8). If post-bariatric surgery, weight must be stable ±5% (self-report) for at least 6 months prior to first dose of study drug (Day 8).
* Any form of medically managed weight loss program within 6 months prior to the first dose of study drug (Day 8);
* Significant defect in nasal patency due to anatomical abnormalities or uncontrolled or recurrent episodes of rhinitis;
* Any clinically significant unstable or progressive medical condition;
* Any primary sleep disorder other than OSAS as determined by history, physical examination, or Visit 2 PSG (after 7-day screening run-in period);
* Clinically significant or uncontrolled: chronic obstructive pulmonary disease (COPD), cardiovascular disease, gastrointestinal, respiratory, pancreatic, hepatic, renal, hematologic, endocrine [including insulin-dependent diabetes mellitus (IDDM)], neurological, urogenital, connective tissue, dermatological, thyroid, or other medical disorder;
* Any clinically significant psychiatric disorder;
* History of seizure disorder;
* Treatment with any prescription antidepressant medication within 1 month prior to the first dose of study drug (Day 8);
* Treatment with sedatives, hypnotics or other psychoactive drugs within 30 days prior to the first dose of study drug (Day 8);
* Any complete blood count (CBC) or liver function test (LFT) laboratory value outside the normal range which, in the clinical judgment of the Investigator renders a subject inappropriate for randomization to treatment;
* Pregnancy [as demonstrated by positive urine human chorionic gonadotropin (hCG) test] or lactation;
* Allergic to cannabinoids or sesame oil;
* History of substance abuse (including alcohol abuse or dependence) or laboratory evidence of drug abuse on the Visit 1 drug-screening panel;
* Use of dietary supplements which in the judgment of the Investigator may impact sleep or breathing behaviors;
* Average daily caffeine consumption > 500 mg/day (~5 cups of coffee);
* Average weekly alcohol consumption > 10 units;
* Unwillingness to abstain from caffeine and alcohol on all days when overnight or daytime testing will be performed;
* Participation in any other investigational protocol within the 30 days prior to the first dose of study drug (Day 8);
* Any condition which, in the opinion of the Investigator, places the patient at unacceptable risk if he or she were to participate in the study.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2013-02; Primary Completion 2016-06 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David W Carley, PhD, Principal Investigator — University of Illinois at Chicago
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois

REFERENCES:
- [Derived] Carley DW, Prasad B, Reid KJ, Malkani R, Attarian H, Abbott SM, Vern B, Xie H, Yuan C, Zee PC. Pharmacotherapy of Apnea by Cannabimimetic Enhancement, the PACE Clinical Trial: Effects of Dronabinol in Obstructive Sleep Apnea. Sleep. 2018 Jan 1;41(1):zsx184. doi: 10.1093/sleep/zsx184. PMID 29121334

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from physician referrals at two academic medical centers as well as from the community based upon print and radio advertising between January 2013 and May 2016. The first participant was enrolled in February 2013 and the last participant was enrolled in April 2016.
Groups:
- Sugar Pill: Placebo, once per day (QD) by mouth, 60 minutes before bedtime for 6 weeks after 1-week run-in
  Placebo (for Dronabinol)
- 2.5 mg/Day: Dronabinol, 2.5 mg QD by mouth, 60 minutes before bedtime for 6 weeks after 1-week placebo run-in
  Dronabinol
- 10 mg/Day: Dronabinol, 10 mg QD by mouth, 60 minutes before bedtime for 4 weeks after 1-week placebo run-in and 2-week dose escalation
  Dronabinol
Period: Overall Study
Arm/Group | Sugar Pill | 2.5 mg/Day | 10 mg/Day
Started | 26 | 22 | 27
Completed | 17 | 19 | 20
Not Completed | 9 | 3 | 7
Not completed — Withdrawal by Subject | 6 | 1 | 3
Not completed — Adverse Event | 1 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Physician Decision | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Baseline analysis population includes all participants who were randomized to treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugar Pill | 2.5 mg/Day | 10 mg/Day | Total
Number analyzed (Participants) | 26 | 22 | 27 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 26 | 22 | 27 | 75
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 9 | 23
  Male | 18 | 16 | 18 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 1 | 10
  Not Hispanic or Latino | 22 | 17 | 25 | 64
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 15 | 5 | 13 | 33
  White | 9 | 16 | 12 | 37
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 33.39 (6.33) | 33.19 (5.09) | 33.45 (4.85) | 33.35 (6.33)
Apnea/Hypopnea Index [Mean (Standard Deviation); unit: events/hour] | 23.72 (9.47) | 27.54 (12.57) | 26.04 (11.92) | 25.67 (11.29)
Minimum Arterial Oxygen Saturation [Mean (Standard Deviation); unit: %] | 79.58 (9.62) | 79.82 (6.83) | 79.96 (6.93) | 79.79 (7.84)
Sleep Efficiency [Mean (Standard Deviation); unit: %] — Sleep Efficiency is calculated as the total time spent asleep divided by the total amount of time spent in bed, multiplied by 100.
  % | 75.51 (12.50) | 80.52 (11.11) | 82.74 (12.22) | 79.58 (12.25)

OUTCOME MEASURES:

1. Primary Outcome: Change in Apnea/Hypopnea Index (AHI)
Description: Change in AHI derived as: AHI (end of treatment) minus AHI (pre-treatment)
Time Frame: Baseline and Week 6
Population: Analysis performed including all participants who completed the full 6-weeks of treatment.
Measure: Mean (Standard Deviation); unit: events/hour
Arm/Group | Sugar Pill | 2.5 mg/Day | 10 mg/Day
Number analyzed (Participants) | 17 | 19 | 20
events/hour | 7.99 (13.16) | -1.71 (11.74) | -5.21 (9.52)

2. Primary Outcome: Change in Epworth Sleepiness Scale (ESS)
Description: Change in ESS derived as: ESS (end of treatment) minus ESS (pre-treatment). The ESS scale has a range of 0 to 24, with 0 representing the least degree of sleepiness and 24 the greatest degree of sleepiness. There are no subscales.
Time Frame: Baseline and Week 6
Population: Data are missing for 2 participants randomized to receive Placebo treatment; due to technical error in not completing this instrument.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sugar Pill | 2.5 mg/Day | 10 mg/Day
Number analyzed (Participants) | 15 | 19 | 20
units on a scale | -1.47 (3.29) | -.26 (2.94) | -4.00 (5.13)

3. Primary Outcome: Change in Sleep Latency: Maintenance of Wakefulness Test (MWT)
Description: Change in MWT derived as: MWT (end of treatment) minus MWT (pre-treatment). The Maintenance of Wakefulness Test measures a person's ability to stay awake in a quiet, dark and nonstimulating room for a period of time.
Time Frame: Baseline and Week 6
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sugar Pill | 2.5 mg/Day | 10 mg/Day
Number analyzed (Participants) | 17 | 19 | 20
minutes | -2.50 (13.09) | -3.70 (9.73) | 1.40 (11.71)

4. Secondary Outcome: Tolerability by Treatment Satisfaction Questionnaire for Medications (TSQM) Overall Score.
Description: The TSQM measures a person's satisfaction with treatment based on a 7-point scale ranging from "Extremely Dissatisfied" to "Extremely Satisfied" in response to the question, "Taking all things into account, how satisfied or dissatisfied are you with this medication?".
Time Frame: Week 6
Population: Data are missing for one participant randomized to receive Placebo treatment due to technical error in not collecting the instrument.
Measure: Count of Participants; unit: Participants
Arm/Group | Sugar Pill | 2.5 mg/Day | 10 mg/Day
Number analyzed (Participants) | 16 | 19 | 20
Participants
  Extremely Dissatisfied | 3 | 2 | 1
  Very Dissatisfied | 1 | 2 | 0
  Dissatisfied | 0 | 3 | 0
  Somewhat Satisfied | 5 | 6 | 4
  Satisfied | 1 | 4 | 4
  Very Satisfied | 5 | 1 | 5
  Extremely Satisfied | 1 | 1 | 6

5. Secondary Outcome: Adverse Events (AEs)
Description: AEs will be evaluated and tracked throughout subject participation (up to 8 weeks)
Time Frame: Up to 8 weeks
Measure: Mean (Standard Deviation); unit: Number of adverse events per participant
Arm/Group | Sugar Pill | 2.5 mg/Day | 10 mg/Day
Number analyzed (Participants) | 26 | 22 | 27
Number of adverse events per participant | 3.4 (2.9) | 2.8 (3.6) | 5.8 (4.7)

6. Secondary Outcome: Change in Desaturation Time (DT)
Description: Change in DT (total minutes with arterial oxygen saturation below 85% during 8-hour polysomnography) derived as: DT (end of treatment) minus DT (pre-treatment)
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sugar Pill | 2.5 mg/Day | 10 mg/Day
Number analyzed (Participants) | 17 | 19 | 20
minutes | 1.21 (3.46) | -0.19 (2.78) | -0.17 (6.68)

ADVERSE EVENTS:
Arm/Group | Sugar Pill | 2.5 mg/Day | 10 mg/Day
Serious Adverse Events (participants affected / at risk) | 1/26 | 1/22 | 0/27
Other Adverse Events (participants affected / at risk) | 9/26 | 13/22 | 26/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugar Pill (N=26) | 2.5 mg/Day (N=22) | 10 mg/Day (N=27)
Cycling injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Struck by vehicle while riding a bicycle
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugar Pill (N=26) | 2.5 mg/Day (N=22) | 10 mg/Day (N=27)
Sleepy (Nervous system disorders) | 0 (0) | 0 (0) | 17 (17) — Increased sleepiness, tiredness or drowsiness
Diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 4 (4)
Headache (Nervous system disorders) | 4 (4) | 3 (3) | 13 (13)
Nausea (Gastrointestinal disorders) | 1 (1) | 5 (5) | 9 (9) — Nausea or vomiting
Dizziness (Nervous system disorders) | 3 (3) | 1 (1) | 7 (7) — Dizziness or lightheadedness
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Muscle aches (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Euphoria (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) — Euphoria or feeling "high"

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No